CLINICAL TRIAL: NCT06674564
Title: Effect of Zinc and Probiotics Supplementation on Laryngeal Cancer Patients Undergoing Laryngectomy Surgery
Brief Title: Effect of Zinc and Probiotics Supplementation on Laryngeal Cancer Patients Undergoing Laryngectomy Surgery to Improve Prognosis and Better Wound Healing
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: zn probiotics laryngeal cancer
Record Dates: First submitted 2024-10-01; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-09

CONDITIONS: Laryngectomy
Keywords: laryngeal cancer , zinc , probiotics, total laryngectomy
MeSH Terms: conditions — Laryngeal Neoplasms | interventions — Zinc Acetate; Probiotics

STUDY DESIGN:
Intervention Model Description: Model Description
Masking Description: open labelled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- control group (No Intervention): patients in this group will not having any interventions except the usual treatment before and after surgery
- zinc group (Active Comparator): patients in this group will take 50 mg zinc sulfate beside the usual treatment
  Interventions: Dietary Supplement: Zinc Acetate 50 Mg Oral Capsule
- probiotics group (Active Comparator): patients in this group will take probiotics beside the usual treatment
  Interventions: Dietary Supplement: Probiotic
- zinc and probiotics proup (Active Comparator): patients in this group will take zinc and probiotics beside the usual treatment
  Interventions: Dietary Supplement: Zinc Acetate 50 Mg Oral Capsule; Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Zinc Acetate 50 Mg Oral Capsule — zinc suppose to improve immunity and wound healing after laryngectomy
  Arms: zinc and probiotics proup; zinc group
Dietary Supplement: Probiotic — probiotics lowering infections rates and improving outcomes after surgery
  Arms: probiotics group; zinc and probiotics proup

SUMMARY:
using zinc and probiotics supplementation for providing better prognosis for laryngeal cancer patients under going total or partial laryngectomy.

DETAILED DESCRIPTION:
Zinc supplementation decrease plasma levels of oxidative stress markers, inflammatory cytokines and IL6. Low Serum zinc level was believed to influence the survival of laryngeal cancer patients and hence,using zinc supplementation would improve survival.Zinc help in increasing wound healing as involve in membrane repair, decreasing oxidative stress , coagulation , suppressing inflammation and modulating .Probiotics stimulates epithelial cells to release interleukin 6 (IL-6) and stimulates dendritic cells and macrophages that help in releasing TNF-α and IFN-γ , development IgA B lymphocytes that cause increase production of IgM, IgG and IgE antibodies.using probiotics preoperative or post-operative offer good chance for decreasing morbidity , infection rates , abuse of antibiotics and complications. zinc and probiotic suppose to provide better wound healing low incidence of infections and fistula after total and partial laryngectomy

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting to ENT department will be subjected eligible Adults patients newly diagnosed at outpatient clinic with laryngeal cancer at any stage and will undergo total/partial laryngectomy surgery.

Patients with Level of hemoglobin >9 mg/dl and serum albumin 3g/dl According to (Crosetti et al. 2021).

Staging of laryngeal cancer according to the American Joint Committee on Cancer (AJCC) 8th edition by TNM system.

Exclusion Criteria:

- 1. Impaired renal function sr.cr≤2.5 (zinc clearance). 2.Previous history of cancer diseases in other sites( previous chemotherapy or radiation).

3.Hypersensitivity to probiotics and zinc.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2024-09-09 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
wound healing | 21 days after surgery, a month total
  The role of zinc and probiotics supplementations on the rate of wound healing (pharyngeal reconstruction.
occurrence of percutaneous fistula | 21 days after surgery - total a month
  according to john et al grading 3- 4 grade
rate of infections | 21 days after surgery - a month total
  rate of infection of wound after total /partial laryngectomy
starting of oral feeding | 21 days after surgery-30 days total
  reconstruction of pharynx post operative and start oral feeding

SECONDARY OUTCOMES:
length of hospital stay | month from start , 21 days after surgery
  length of hospital stay (hospital discharge)
evaluation of safety of probiotics and zinc supplementations in adults patients after total/ partial laryngectomy in terms of adverse drug events. | 21-days post surgery month total
  evaluation of safety of probiotics and zinc supplementations in adults patients after total/ partial laryngectomy in terms of adverse drug events.

CONTACTS AND LOCATIONS:
Overall Officials: botamina nabil, Principal Investigator — pharmacy ASU
Locations (1):
- Ain shams university hospital, Cairo, Al Abbasya, Egypt

IPD SHARING:
Plan to Share IPD: No
until the reaserch would be complete